CLINICAL TRIAL: NCT00498420
Title: A Multicenter, Multinational Study That Will Evaluate Clinical and Surrogate Parameters Known to be Affected in Alpha-Mannosidosis Patients
Brief Title: The Natural History of Alpha-Mannosidosis
Acronym: HUE-MAN
Status: Completed | Type: Observational
Sponsor: Zymenex A/S (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Other Study IDs: rhLAMAN-01; 2004-2.1.1-10
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Alpha Mannosidosis
Keywords: HUE-MAN; Rare disorder; Hepatosplenomegaly; Dysostosis
MeSH Terms: conditions — alpha-Mannosidosis; Rare Diseases; Dysostoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The natural history study of the rare lysosomal disease alpha-mannosidosis will answer the question; why the rare disease develops as it does?

DETAILED DESCRIPTION:
Definition:

Human alpha-mannosidosis is a rare genetic disorder, caused by the lack of lysosomal alpha-mannosidase, resulting in mental retardation, skeletal changes, hearing loss and recurrent infections. The lack of alpha-mannosidase causes a disorder of glycoprotein catabolism associated with abnormal levels and excretion of small mannose-rich oligosaccharides.

Prevalence:

Alpha-mannosidosis belongs to a group of lysosomal storage disorders that includes more than 50 different diseases, with a cumulative frequency of about 1:10.000 world wide. The incidence of alpha-mannosidase disease has been estimated to be 1 in 500.000 (Australian and Norwegian study). The disease is not specific to any ethnic group.

Etiology and Pathogenesis:

Lysosomal alpha-mannosidase (LAMAN), in the following called mannosidase, is an enzyme that cleaves alpha-mannosidic linkages during the ordered degradation of oligosaccharides. Only after degradation, can the sugars leave the lysosomes, the cell and later the body. The deficiency in mannosidase activity causes a block in the degradation of glycoproteins resulting in lysosomal accumulation of mannose-rich oligosaccharide chains. Consequently, these sugars accumulate in the lysosomes as they are too large to leave. Finally, the lysosomes increase in size, producing vacuoles and impaired cellular function is induced by an unknown mechanism.

Clinical Findings:

Affected children are usually born apparently normal and their condition worsens progressively without any possible treatment available to prevent this evolution. The clinical findings in alpha-mannosidosis include a broad range of symptoms, from an early lethal form to less symptomatic, chronic forms often initially diagnosed in childhood. Alpha-mannosidosis is frequently associated with corneal opacities, aseptic destructive arthritis, metabolic myopathy and immune deficiency. In the past alpha-mannosidosis was classified into two forms. A more severe infantile (type 1) phenotype that include rapid, progressive mental retardation; hepatosplenomegaly; severe dysostosis multiplex; and often death between 3 and 12 years of age. The juvenile-adult phenotype (type 2) is characterized by a milder and more slowly progressive course with survival into adulthood. The distinctions are not absolute, and symptoms and lethality may vary. In affected children that are born healthy, there is a window of opportunity for a therapy initiated at an early age to contribute to normal development and the prevention of other disease related complications.

Study objectives:

To assess the short-term, natural history of subjects diagnosed with Alpha-Mannosidosis To establish the range and diversity of clinical symptomatology To evaluate short term (24 months) changes in disease parameters

ELIGIBILITY:
Inclusion Criteria:

1. The patient (or patient's legal guardian) must provide written informed consent prior to performing any survey-related procedures.
2. The patient must have a documented diagnosis of Alpha Mannosidosis, confirmed at screening by measurable clinical signs and symptoms of Alpha Mannosidosis
3. Documented deficiency of serum or leukocyte acid alpha-mannosidase enzyme activity level

Exclusion Criteria:

1. History of bone marrow transplantation.
2. Use of an investigational drug within 30 days prior to study enrollment.
3. Known medical condition, serious intercurrent illness, or other extenuating circumstance that may significantly decrease study compliance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: To be eligible to proceed, each subject must meet all inclusion and exclusion criteria during the screening periode.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-05; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Beck, MD, Principal Investigator — Children's Hospital, University of Mainz; Ed Wraith, MD, Principal Investigator — Willink Biochemical Genetics Unit, Royal Manchester Childern's Hospital; Jiri Zeman, MD, Principal Investigator — Department of Pediatrics, Charles University; Dag Malm, MD, Principal Investigator — Department of Medicine, University of Tromsoe
Locations (4):
- Department of Pediatrics, Charles University, Prague, Czechia
- University of Mainz, Mainz, Germany
- Department of Medicine, University of Tromsoe, Tromsø, Norway
- Willink Biochemical Genetics Unit,. Royal Manchester Children's Hospital, Manchester, United Kingdom

REFERENCES:
- [Result] Beck M, Olsen KJ, Wraith JE, Zeman J, Michalski JC, Saftig P, Fogh J, Malm D. Natural history of alpha mannosidosis a longitudinal study. Orphanet J Rare Dis. 2013 Jun 20;8:88. doi: 10.1186/1750-1172-8-88. PMID 23786919
- [Result] Borgwardt L, Stensland HM, Olsen KJ, Wibrand F, Klenow HB, Beck M, Amraoui Y, Arash L, Fogh J, Nilssen O, Dali CI, Lund AM. Alpha-mannosidosis: correlation between phenotype, genotype and mutant MAN2B1 subcellular localisation. Orphanet J Rare Dis. 2015 Jun 6;10:70. doi: 10.1186/s13023-015-0286-x. PMID 26048034
- See also: These websites are dedicated to the HUE-MAN project — http://www.uni-kiel.de/Biochemie/hue-man/index.htm